CLINICAL TRIAL: NCT02298920
Title: A Phase I, Open-Label Study to Assess the Absorption, Metabolism, Excretion, Safety and Tolerability of a Single Oral Dose of Radiolabeled [14C]-AZD0914 in Healthy Male Subjects
Brief Title: AZD0914 Phase 1 ADME Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4930C00003
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — zoliflodacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group (Experimental): Open Label ADME Study
  Interventions: Drug: AZD0914

INTERVENTIONS:
Drug: AZD0914 — Radiolabelled AZD0914 for study of absorption, disposition, metabolism, and excretion in healthy volunteers.

SUMMARY:
This study will investigate the metabolic fate and routes of excretion of 14CAZD0914 in six male healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, single dose study in 6 healthy male subjects aged 18 to 55 years. Each subject will be admitted to the clinical pharmacology unit on the day prior to dosing Check in (Day -1) and will remain in the clinical pharmacology unit until up to at least target Day 8 (168 hours post-dose).

All subjects will receive 3000 mg AZD0914 incorporating 18.5 MBq (500 Ci) of [14C] administered as a single oral dose following at least an 8 hour fast from food. Subjects can have water. For specific food and water restrictions.

This study will investigate the metabolic fate and routes of excretion of AZD0914.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18 and 55 years of age, inclusive, at the time of consent with suitable veins for cannulation or repeated venipuncture;
2. Subjects must be able to understand and be willing to comply with study procedures, restrictions, and requirements;
3. Within body mass index (BMI) range 19 to 30 kg/m2, inclusive, at screening;
4. Non-smokers in past 6 months;
5. In good health, as determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs as judged by the Investigator;

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, interfere with absorption, distribution, metabolism or excretion of drugs, or influence the results or the subject's ability to participate in the study;
2. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QT interval corrected for heart rate (QTc) changes;
3. Any clinically significant abnormalities in clinical chemistry, hematology, or UA results as judged by the Investigator;
4. Abnormal vital signs, after 10 minutes supine rest, confirmed by repeat, defined as any of the following: systolic blood pressure <90 mmHg or >140 mmHg; diastolic blood pressure <50 mmHg or >90 mmHg; or heart rate <40 or >100 beats per minute;
5. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IP;

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PK Parameters | Up to 11 days
  Maximum observed concentration (Cmax), time to maximum observed concentration (tmax), area under the concentration-time curve from hour 0 to the last measurable concentration (AUC0-t), area under the concentration-time curve extrapolated to infinity (AUC0-inf), apparent terminal elimination rate constant (lambdaZ), apparent terminal elimination half-life (t1/2), apparent clearance (Cl/F) (oral and AZD0914 only), and apparent volume of distribution (Vz/F) (AZD0914 only). Ratios for area under the concentration-time curve extrapolated to infinity including the ratio of total radioactivity in whole blood/plasma and the ratio of non-radiolabeled AZD0914 in plasma/total radioactivity in plasma, will be calculated as appropriate.
Urine and Feces PK Parameters | Up to 11 days
  The following pharmacokinetic parameters will be calculated, whenever possible, based on the urine total radioactivity concentrations: amount excreted in urine (Aeu) over the sampling interval, renal clearance (CLR), and the percent excreted in urine (%Feu). For fecal total radioactivity concentrations, the following pharmacokinetic parameters will be calculated for [14C] AZD0914 derived radioactivity: amount excreted in feces (Aef) over the sampling interval and the percent excreted in feces (%Fef).
Metabolites | Up to 11 days
  Metabolites of [14C]-AZD0914 will be identified. Pharmacokinetic parameters for the metabolites of [14C]-AZD0914 will be calculated, as deemed appropriate, based on plasma and urine concentration levels. Data may be presented in a separate report.

SECONDARY OUTCOMES:
Number and severity of adverse events, abnormal labs, signs, ECGs, and PEs | Up to 17 days
  Signs, symptoms, incidence, and severity of adverse events (AE), abnormalities in clinical laboratory assessments, vital signs, electrocardiograms (ECGs), and physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Mirkin, MD, Principal Investigator — Covance Clinical Research Unit
Locations (2):
- United States (2):
  - Covance Clinical Research Unit, Madison, Wisconsin
  - Research Site, Madison, Wisconsin

REFERENCES:
- [Derived] O'Donnell J, Lawrence K, Vishwanathan K, Hosagrahara V, Mueller JP. Single-Dose Pharmacokinetics, Excretion, and Metabolism of Zoliflodacin, a Novel Spiropyrimidinetrione Antibiotic, in Healthy Volunteers. Antimicrob Agents Chemother. 2018 Dec 21;63(1):e01808-18. doi: 10.1128/AAC.01808-18. Print 2019 Jan. PMID 30373802